CLINICAL TRIAL: NCT03741413
Title: Saving a Life or Preventing a Death: the Effect of Message Framing on Blood Donation Among Rh Negative Donors
Brief Title: The Effect of Message Framing on Blood Donation-Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Blood Center (Other Government)
Responsible Party: Principal Investigator, OUYANG Jian, MS, Guangzhou Blood Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Message framing effect
Record Dates: First submitted 2018-11-11; First posted 2018-11-14 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Rh Negative Blood Donor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Gain-frame SMS (Experimental): SMS messages "Dear Rh negative blood donors: Hello! As the Rh negative O/B blood stockpile is low now, but patients who are this blood type are in urgent need. If you are available, we hope that you can offer a helping hand to save their lives. Thank you for your support." were send to donors in this group.
  Interventions: Other: Gain-frame SMS
- Loss-frame SMS (Experimental): SMS messages "Dear Rh negative blood donors: Hello! As the Rh negative O/B blood stockpile is low now, but patients who are this blood type are in urgent need. If you are available, we hope that you can offer a helping hand to prevent them from death. Thank you for your support." were send to donors in this group.
  Interventions: Other: Loss-frame SMS
- Control SMS (Experimental): SMS messages "Dear Rh negative blood donors: Hello! As the Rh negative O/B blood stockpile is low now, but patients who are this blood type are in urgent need. If you are available, we hope that you can donate blood again. Thank you for your support." were send to donors in this group.
  Interventions: Other: Control SMS
- Control group (No Intervention): Donors in this group were not received SMS reminders.

INTERVENTIONS:
Other: Gain-frame SMS — Emergency recruitment cell phone short messages that emphasizing donating blood can save patients' lives were sent to donors in this group.
  Arms: Gain-frame SMS
Other: Loss-frame SMS — Emergency recruitment cell phone short messages emphasizing that donating blood can prevent patients from death were sent to donors in this group.
  Arms: Loss-frame SMS
Other: Control SMS — Emergency recruitment cell phone short messages that only mentioning the low Rh-negative blood stockpile were sent to donors in this group.
  Arms: Control SMS

SUMMARY:
Rh negative blood group is a rare blood group in China, as it only accounts for 0.3-0.4 percent of the Han population. Therefore, low inventory is often found in blood collection and supply agencies in many regions in China. On July 18, 2018 blood stockpile of O-negative and B-negative in Guangzhou Blood Center reached the warning line, and we took measures for emergency recruitment. O-negative and B-negative blood donors whose last donation dates were between January 1, 2015 and December 31, 2017 were identified and randomly assigned to three groups. Three different recruitment text messages were send to these groups respectively. At the same time, A-negative and AB-negative blood donors were marked as control group. We observed the re-donation rates among four groups within three months.

ELIGIBILITY:
Inclusion Criteria:

* Rh- negative blood donors whose last donations were between January 1, 2015 and December 31, 2017.

Exclusion Criteria:

* Donors with an obviously invalid phone number. Donors whose serological results of the last donation were positive.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2074 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Re-donation rate | 3 months
  Intention-to-treat were applied. Re-donation rate was defined as the number of donors in each group devided by donors who re-donated within 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Blood Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No